CLINICAL TRIAL: NCT06927245
Title: Use of Intraoperative Autofluorescence Imaging to Reduce the Incidence of Inadvertent Parathyroidectomy During Thyroid Surgery
Brief Title: Use of the PTEye Device to Reduce Inadvertent Parathyroidectomy During Thyroid Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProMedica Health System (Other)
Responsible Party: Principal Investigator, Joseph Sferra, Professor, Department of Surgery, ProMedica Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Record Dates: First submitted 2025-03-10; First posted 2025-04-15 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-04

CONDITIONS: Thyroid Surgery; Inadvertent Parathyroidectomy; Enlarged Thyroid
Keywords: PTEye; Total Thyroidectomy; Thyroid Lobectomy; Intraoperative Autofluorescence Imaging; Inadvertent Parathyroidectomy; Inadvertent Parathyroid Removal
MeSH Terms: conditions — Goiter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients receiving Thyroid Surgery (Experimental): The experimental treatment group that is having either a Total Thyroidectomy or a Thyroid Lobectomy procedure done will have the PTEye device used in surgery to identify their Parathyroid Gland through autofluorescence.
  Interventions: Device: PTeye Device

INTERVENTIONS:
Device: PTeye Device — Near infrared stimulation of parathyroid tissue using light at a wavelength of approximately 690 - 770 nm results in autofluorescence of parathyroid tissue. Near infrared autofluorescence detection devices, such as PTEye have been developed with probe-based methods, displaying quantitative real-time information to aid surgeons in detection of parathyroid tissue relative to surrounding tissue.
  Other Names: Intraoperative Autofluorescence Imaging

SUMMARY:
Inadvertent Parathyroidectomy (IP) during thyroid surgery may lead to transient or permanent hypoparathyroidism and hypocalcemia, which represents significant morbidity. Patients that suffer from IP and its clinical consequences often require longer duration of hospitalization and additional inpatient treatment and prescription medications. ProMedica performs a large number of endocrine procedures, so the use of novel technology to aid in the intra operative identification of parathyroid glands may ultimately offer decreased morbidity to patients.

The goal of this study is to find out if using the PTEye device (a device that uses infrared light to find the Parathyroid gland) lowers the amount of times a surgeon accidentally takes out the Parathyroid gland while trying to take out the Thyroid gland in surgery.

DETAILED DESCRIPTION:
Inadvertent Parathyroidectomy (IP) during thyroid surgery may lead to transient or permanent hypoparathyroidism and hypocalcemia, which represents significant morbidity. Patients that suffer from IP and its clinical consequences often require longer duration of hospitalization and additional inpatient treatment and prescription medications. ProMedica performs a large number of endocrine procedures, so the use of novel technology to aid in the intra operative identification of parathyroid glands may ultimately offer decreased morbidity to patients.

The investigators plan to prospectively enroll 25 patients undergoing either thyroid lobectomy or total thyroidectomy. The surgeries will be performed by study approved surgeons. All surgeries will take place over a 90 day period beginning at the receipt of the PTEye device. All subjects will be consented pre-operatively for enrollment in the study, including consent for use of the PTeye device. Subjects undergoing a planned parathyroidectomy, Cistrunk procedure, repeat neck surgery, or neck dissection will not be included in this particular study.

Subjects will not have any changes in their pre-surgical procedure. Subjects will follow typical standard of care procedures for surgery. Once the subject is in surgery, the surgeon will use the PTeye device to identify the parathyroid gland. Using the disposable probe to make contact with the tissue, the surgeon will scan the thyroid for a baseline reading. Once the surgeon has established a baseline, they are able to use the device to confirm whether the tissue they identified is parathyroid tissue. The device will make a noise when it detects parathyroid tissue. Other than the use of the PTeye device, the surgeons will follow standard of care procedures to perform the surgery. The subject will follow standard of care post-operative procedures and will not be required to attend any additional appointments (other than those scheduled per standard of care).

The investigators will extract multiple data points from these 25 subjects. The primary endpoint will be the rate of inadvertent parathyroidectomy. This will be identified by review of surgical pathology reports for parathyroid tissue. Secondary endpoints include the number of frozen sections sent, number of autotransplantations of parathyroid tissue performed, operative times, and post operative Parathyroid Hormone and Calcium levels. These data points will be collected by chart review. Each subject will follow up two weeks post operatively, per standard of care procedure. We plan to follow patients for one month post operatively to monitor for any pertinent hospital readmissions by performing a chart review of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing either a total thyroidectomy or a thyroid lobectomy
* Patients must be 18 years old or older
* Patient needs to be operated on by a study approved surgeon

Exclusion Criteria:

* Under 18 years old
* Receiving a planned parathyroidectomy, Cistrunk procedure, repeat neck surgery, or neck dissection
* Receiving surgery from a non-approved surgeon
* Pregnant at time of procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Inadvertent Parathyroidectomy | From enrollment to one month after surgery
  The aim of this study is to establish the rate of inadvertent parathyroidectomy during thyroid surgery when the PTeye near-infrared device is used to aid with intraoperative identification of the parathyroid gland.

IPD SHARING:
Plan to Share IPD: No